CLINICAL TRIAL: NCT03539731
Title: A Phase I Study of [18F]DASA-23 as a PET Tracer for Evaluating Pyruvate Kinase M2 (PKM2) Expression in Healthy Volunteers and in Patients With Intracranial Tumors
Brief Title: [18F]DASA-23 and PET Scan in Evaluating Pyruvate Kinase M2 Expression in Patients With Intracranial Tumors or Recurrent Glioblastoma and Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study did not meet its objectives due to difficulties in enrollment
Sponsor: Guido A. Davidzon, MD, SM (Other)
Responsible Party: Sponsor-Investigator, Guido A. Davidzon, MD, SM, Clinical Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-44597; NCI-2018-00826 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 44597 (Other: Stanford IRB)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subject; Intracranial Neoplasm; Glioblastoma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I ([18F]DASA-23, PET) (Active Comparator): Healthy volunteers receive [18F]DASA-23 IV and undergo brain PET scan over 15 minutes and 4 vertex-to-toe PET scans over 30 minutes each.
  Interventions: Drug: Fluorine F 18 DASA-23; Procedure: Positron Emission Tomography
- Group II ([18F]DASA-23, PET) (Experimental): Intracranial tumor participants receive [18F]DASA-23 IV and undergo brain PET scan over 60 minutes and 1 vertex-to-toe PET scan over 30 minutes.
  Interventions: Drug: Fluorine F 18 DASA-23; Procedure: Positron Emission Tomography
- Group III ([18F]DASA-23, PET) (Experimental): Patients with at least a 1cm3 contrast-enhancing lesion suspicious for GBM (either newly-diagnosed or 1st /2nd/ 3rd recurrence of GBM) on a standard-of-care (SOC) brain MRI scan. If the patient undergoes a biopsy or resection for GBM (either newly-diagnosed or 1st /2nd/ 3rd recurrence of GBM) then the remaining contrast-enhancing lesion is at least 1cm3 in size on the post-operative scan. These patients will undergo one [18F]DASA 23 PET/MRI scan before the initiation of therapy, and a second/final [18F]DASA 23 PET/MRI scan within 2-6 weeks after initiation of therapy for their GBM.
  Interventions: Drug: Fluorine F 18 DASA-23; Procedure: Positron Emission Tomography
- Group IV ([18F]DASA-23, PET) (Active Comparator): Healthy volunteers receive [18F]DASA-23 IV and undergo brain PET/MRI brain scan for 60 mins
  Interventions: Drug: Fluorine F 18 DASA-23; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Fluorine F 18 DASA-23 — Given IV
  Other Names: [18F]DASA-23; [18F]DASA23; 18F-DASA-23; 1-((2-Fluoro-6-[18F]fluorophenyl)sulfonyl)-4-((4-methoxyphenyl)sulfonyl)piperazine; F18-labeled Pyruvate Kinase M2 Inhibitor DASA-23; F18-labeled PKM2 Inhibitor
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I trial studies how well [18F]DASA-23 and positron emission tomography (PET) scan work in evaluating pyruvate kinase M2 (PKM2) expression in patients with intracranial tumors or recurrent glioblastoma and healthy volunteers. PKM2 regulates brain tumor metabolism, a key factor in glioblastoma growth. [18F]DASA-23 is a radioactive substance with the ability to monitor PKM2 activity. A PET scan is a procedure in which a small amount of a radioactive substance, such as [18F]DASA-23, is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the substance is used. Tumor cells usually pick up more of these radioactive substances, allowing them to be found. Giving [18F]DASA-23 with a PET scan may help doctors evaluate PKM2 expression in healthy volunteers and in participants with intracranial tumors or recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the fluorine F 18 DASA-23 ([18F]DASA 23) PET scan signal change from pre-therapy to one week after initiation of therapy can predict the tumor's responsiveness to therapy and 6 month progression free survival (PFS6), in suspected recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. Determine the sensitivity, specificity, and accuracy of [18F]DASA-23 PET imaging in identifying intracranial tumors in patients with intracranial tumors.

II. Determine whether the [18F]DASA-23 PET scan signal change from pre therapy to one week after initiation of therapy can predict progression free survival (PFS) and overall survival (OS), in suspected recurrent glioblastoma.

OUTLINE: Participants are assigned to 1 of 4 groups.

GROUP I: Healthy volunteers receive [18F]DASA-23 intravenously (IV) and undergo brain PET scan over 15 minutes and 4 vertex-to-toe PET scans over 30 minutes each.

GROUP II: Intracranial tumor participants receive [18F]DASA-23 IV and undergo brain PET scan over 60 minutes and 1 vertex-to-toe PET scan over 30 minutes.

GROUP III: Subjects with glioblastoma will receive [18F]DASA-23 IV and undergo brain PET scan over 60 minutes and 1 vertex-to-toe PET scan over 30 minutes. 15-minute vertex-to-thigh PET for Part 3 patients, Participants undergo second PET scan 7 days after the initiation of therapy.

GROUP IV: Healthy volunteers will undergo the same procedures as the healthy volunteers in Group I with the following exceptions:

Group IV healthy volunteers will undergo a 60-minute PET/MRI brain scan instead of a 15-minute PET/MRI brain scan.

Group IV healthy volunteers will not undergo any vertex-to-toe PET scans.

After completion of study treatment, intracranial tumor and recurrent glioblastoma participants are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old.

2. Adequate organ function (obtained within 14 days prior to PET scan [Part 1, Part 2, and Part 3 ONLY] or within 28 days prior to PET scan [Part 4 ONLY]) as evidenced by:

1. ANC ≥ 1.5 X 10^9/L w/o myeloid growth factor support for 7 d preceding lab assessment
2. Hgb ≥ 9 g/dL (90 g/L); < 9 g/dL (< 90 g/L) is acceptable if Hgb is corrected to ≥ 9 g/dL (90 g/L) as by growth factor or transfusion prior to PET scan
3. Platelet count ≥ 100 X 10^9/L w/o blood transfusions for 7 d preceding lab assessment
4. Bilirubin ≤ 1.5 X ULN except for pts w/ documented history of Gilbert's disease
5. ALT and AST ≤ 2.5 X ULN
6. Alkaline phosphatase (AP) ≤ 3 X ULN
7. Women of childbearing potential (WCBP): negative serum pregnancy test

   3. Ability to stand up and climb two steps with minimal assistance.

   4. Ability to understand and the willingness to sign a written informed consent document.

   5. (Part 2, intracranial tumor patients ONLY) (a) Radiographical or pathological evidence of newly-diagnosed intracranial tumor that is status-pre surgical resection, or (b) Radiographical or pathological evidence of progressive/recurrent intracranial tumor, (c) Question of pseudoprogression vs. true progression on most recent standard-of-care brain MRI, or (d) Evidence on the most recent standard-of-care brain MRI scan of intracranial metastasis/metastases in a patient with known extracranial primary cancer.

   6. (Part 3, GBM patients ONLY) Any patient with at least a 1cm3 contrast-enhancing lesion suspicious for GBM (either newly-diagnosed or 1st /2nd/ 3rd recurrence of GBM, molecular GBM, diffuse astrocytomas with molecular features of GBM, H3K27M midline gliomas, gliosarcomas, or any other WHO Grade IV glioma) on a standard-of-care (SOC) brain MRI scan. If the patient undergoes a biopsy or resection for GBM (either newly-diagnosed or 1st /2nd/ 3rd recurrence of GBM, molecular GBM, diffuse astrocytomas with molecular features of GBM, H3K27M midline gliomas, gliosarcomas, or any other WHO Grade IV glioma) then the remaining contrast-enhancing lesion is at least 1cm3 in size on the post-operative scan.

   7. (Part 3, GBM patients ONLY) Life expectancy of ≥ 6 months.

Exclusion Criteria:

1. Known allergy to adhesive tapes or other skin adhesives used in medical care
2. Subjects with the following co-morbid disease or incurrent illness:

   1. With known cirrhosis diagnosed with Child-Pugh Class A or higher liver disease.
   2. Severe/uncontrolled inter-current illness within the previous 28 days prior to PET scan
   3. Patients who have implantable devices that are contra-indicated for MRI
   4. Bleeding disorder
   5. Any other significant co-morbid conditions that in the opinion of the Investigator would impair study participation or cooperation.
   6. (Healthy volunteers ONLY - Part 1 and Part 4) prior or current malignancy
   7. (Healthy volunteers ONLY - Part 1 and Part 4) known kidney disease
3. Pregnant or nursing participants
4. History of allergic reactions to gadolinium-based MRI contrast agent
5. (Part 2, intracranial tumor patients ONLY) Other chemotherapy (besides what is being used to treat the intracranial tumor)
6. (Part 3, GBM patients ONLY) Has already begun therapy, prior to the first of two [18F]DASA-23 PET/MRI scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in [18F]DASA-23 PET scan signal in patients with suspected recurrent glioblastoma | From pre-treatment to one week after initiation of treatment
  Response to treatment is based on the response assessment in neuro-oncology (RANO) criteria. Each patient will be dichotomized into responding (yes) or not responding (no) to treatment based on RANO criteria. The [18F]DASA-23 PET scan signal will be calculated according to the European Organization for Research and Treatment of Cancer (EORTC) response criteria guidelines and reported as median and range, both for the entire cohort as well as separately for the responder and non-responder subgroups. The Mann-Whitney test of [18F]DASA-23 PET scan signal between responders and non-responders will be performed.

SECONDARY OUTCOMES:
Sensitivity of [18F]DASA-23 PET imaging in identifying intracranial tumors in patients with intracranial tumors. | Time of the [18F]DASA-23 PET scan
  Sensitivity will be reported as a percentage with 95% confidence interval.
Specificity of [18F]DASA-23 PET imaging in identifying intracranial tumors in patients with intracranial tumors. | Time of the [18F]DASA-23 PET scan
  Specificity will be reported as a percentage with 95% confidence interval
Accuracy of [18F]DASA-23 PET imaging in identifying intracranial tumors in patients with intracranial tumors. | Time of the [18F]DASA-23 PET scan
  Accuracy will be reported as a percentage with 95% confidence interval.
Progression-free survival in patients with suspected recurrent glioblastoma | Time from diagnosis up to 1 year
  The percent change in SUV from the pre-treatment [18F]DASA-23 PET scan to the post-treatment [18F]DASA23 PET scan will be calculated. Patients will be divided into two groups based on whether their percent change in SUV is above or below the median. Kaplan-Meier curves for the two groups will be plotted and a log-rank test for difference in progression-free survival will be performed. A Cox proportional-hazards regression of progression-free survival on group will be performed. Progression-free survival will be reported as median survival time, with range.
Overall survival in patients with suspected recurrent glioblastoma | From time of initial diagnosis up to 2 years
  The percent change in SUV from the pre-treatment [18F]DASA-23 PET scan to the post-treatment [18F]DASA23 PET scan will be calculated. Patients will be divided into two groups based on whether their percent change in SUV is above or below the median. Kaplan-Meier curves for the two groups will be plotted and a log-rank test for difference in overall survival will be performed. A Cox proportional-hazards regression of overall survival on group will be performed. Overall survival will be reported as median survival time, with range.

CONTACTS AND LOCATIONS:
Overall Officials: Guido A Davidzon, MD, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Derived] Beinat C, Patel CB, Haywood T, Shen B, Naya L, Gandhi H, Holley D, Khalighi M, Iagaru A, Davidzon G, Gambhir SS. Human biodistribution and radiation dosimetry of [18F]DASA-23, a PET probe targeting pyruvate kinase M2. Eur J Nucl Med Mol Imaging. 2020 Aug;47(9):2123-2130. doi: 10.1007/s00259-020-04687-0. Epub 2020 Jan 15. PMID 31938892
- [Derived] Beinat C, Patel CB, Xie Y, Gambhir SS. Evaluation of Glycolytic Response to Multiple Classes of Anti-glioblastoma Drugs by Noninvasive Measurement of Pyruvate Kinase M2 Using [18F]DASA-23. Mol Imaging Biol. 2020 Feb;22(1):124-133. doi: 10.1007/s11307-019-01353-2. PMID 30989436